CLINICAL TRIAL: NCT06756854
Title: Evaluation of Low-Level Laser Therapy as Adjunctive to the Injectable Platelet-Rich Fibrin in the Management of Patients With Thin Gingival Phenotype.
Brief Title: Low-Level Laser Therapy and Injectable Platelet-Rich Fibrin for Thin Gingival Phenotype.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Alaa Elsayed, periodontist, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P-ME-23-05
Record Dates: First submitted 2024-06-21; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Diseases
Keywords: I-PRF, thin gingival phenotype low level laser
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: group1: received I-PRF alone, and group 2: received I-PRF+LLLT
Who Masked: Participant
Masking Description: I-PRF biologic product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test group: injectable platelet rich fibrin+ low level laser therapy (Active Comparator): patients with thin gingival phenotype (gingival thickness less than 1mm) recieve I-PRF+LLLT radiation just after the injection for 3 sessions with 7 days interval between the sessions.
  Interventions: Other: injecable platelet rich fibrin, and low level laser therapy radiation.
- Control group :I-PRF group (Active Comparator): patients with thin gingival phenotype received I-PRF alone in 3 sessions, with 7 days interval between the sessions.
  Interventions: Biological: Biologic Agent: injectable platelet rich fibrin.

INTERVENTIONS:
Biological: Biologic Agent: injectable platelet rich fibrin. — injection of I-PRF to thin gingival phenotype 3 times with 7 days interval between sessions.
  Other Names: Liquid platelet rich fibrin
  Arms: Control group :I-PRF group
Other: injecable platelet rich fibrin, and low level laser therapy radiation. — injection of I-PRF+ exposure to LLLT to thin gingival phenotype 3 times with 7 days interval between sessions.
  Arms: Test group: injectable platelet rich fibrin+ low level laser therapy

SUMMARY:
Management of thin gingival phenotype using non-surgical methods (injection of liquid platelet rich fibrin and exposure to low level laser therapy

DETAILED DESCRIPTION:
Thin gingival phenotype can lead to recession and root exposure. Liquid prf can be obtained by centrifugion of blood sample on speed 700 rpm for 3 min, then injection of this liquid in the attached gingiva and muco-gingival junction (3 times with 7 days interval) for the first group. The second group will be injected with I-PRF in the same method in addition to exposure to Low Level Laser therapy (after each injection of I-PRF). This method is expected to increase the thickness of the gingiva.

ELIGIBILITY:
Inclusion Criteria:

* free systimatically good oral hygiene gingival thickness less than 1mm

Exclusion Criteria:

* pregnancy or lactation pereiodontitis periodontal surgery orthodontic ttt tooth mobility,bruxism,crowding,missing or supernumerary teeth smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Gingival thickness improvement in millimeters. | 6 months after treatment
  clinical parameter
Keratinized tissue width improvement in millimeters. | 6 months after treatment
  Clinincal parameter.

SECONDARY OUTCOMES:
Improvement of gingival index. | 6 months after treatment
  Clinical parameter.
Improvement of bleeding on probing. | 6 months after treatment
  Clinical parameter.
Improvement of sulcus depth. | 6 months after treatment
  Clinical parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Eldawy, doctor, Principal Investigator — MINDRAY
Locations (1):
- Alaa Elsayed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No